CLINICAL TRIAL: NCT07157111
Title: Perioperative Outcomes for Children With Preoperative Upper Respiratory Tract Infection Symptoms in Elective Non-cardiac Surgery After COVID-19 Pandemic at a Large Tertiary Hospital in China: a Retrospective Cohort Study
Brief Title: Perioperative Outcomes for Children With Preoperative URTI Symptoms After COVID-19 Pandemic
Acronym: URTI
Status: Completed | Type: Observational
Sponsor: aijun xu (Other)
Responsible Party: Sponsor-Investigator, aijun xu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: PPOC
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: URTI; Postoperative Complications; COVID - 19; Elective Non-cardiac Surgery; Perioperative Respiratory Adverse Events
MeSH Terms: conditions — Postoperative Complications; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- S1 group: children with preoperative upper respiratory tract infections symptoms undergoing elective non-cardiac surgery from January 1, 2015, to December 31, 2019
- C1 group: children without preoperative upper respiratory tract infections undergoing elective non-cardiac surgery from January 1, 2015, to December 31, 2019
- S2 group: children with preoperative upper respiratory tract infections symptoms undergoing elective non-cardiac surgery from January 1, 2020, to December 31, 2024
- C2 group: children without preoperative upper respiratory tract infections symptoms undergoing elective non-cardiac surgery from January 1, 2020, to December 31, 2024

SUMMARY:
The goal of this observational study is to investigate the impact of the COVID-19 pandemic on perioperative outcomes in children with preoperative URTI symptoms and to explore whether the COVID-19 pandemic affected the additional surgical risk associated with preoperative URTI symptoms. The main question it aims to answer is the appropriate timing of elective non-cardiac surgery in the post-COVID-19 era.

DETAILED DESCRIPTION:
This study aims to investigate the impact of the COVID-19 pandemic on perioperative outcomes in children with preoperative URTI symptoms and to explore whether the COVID-19 pandemic affected the additional surgical risk associated with preoperative URTI symptoms. The findings will provide evidence-based guidance for optimizing surgical timing decisions in the post-COVID-19 era.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0-12 years
* ASA physical status classification I-III
* Undergoing non-cardiac surgery
* Children presenting with mild URTI symptoms within 2 weeks before surgery

Exclusion Criteria:

* Presenting with severe underlying diseases (e.g., congenital heart disease, immunodeficiency)
* Presenting with a single symptom of fever that can be explained by other diseases
* Day surgery
* Children with abnormal preoperative chest X-rays

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 0-12 years who underwent elective non-cardiac surgery at Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology between January 2015 and December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 2392 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 7days
  The postoperative complications including hemorrhage, infection, gastrointestinal complications, respiratory adverse events (RAE), and recurrence of the primary disease.

SECONDARY OUTCOMES:
Intraoperative RAE | 1day
  Intraoperative RAE, including hypercapnia, hypoxemia
Emergence RAE | 1day
  Emergence RAE, including hypercapnia, hypoxemia
PACU stay | 1hour
  Meeting discharge criteria from PACU
Total hospital length of stay | 10days
  Total hospital length of stay
Postoperative length of stay | 7days
  Postoperative hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: aihua Du, Dr., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
Protecting research participant privacy